CLINICAL TRIAL: NCT01095315
Title: Delayed Positioning in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jung-Won Hwang, Seoul National University Bundan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: delayed positioning
Record Dates: First submitted 2010-03-22; First posted 2010-03-30 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-03

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

ARMS (2):
- standard (No Intervention): parturients were placed back to the supine position immediately after spinal injection following standard protocol of spinal anesthesia
- lateral (Experimental): the lateral position was maintained for 6 min after spinal injection before patients were turned to the supine position
  Interventions: Other: lateral positioning

INTERVENTIONS:
Other: lateral positioning — the lateral position was maintained for 6 min after spinal injection before patients were turned to the supine position
  Arms: lateral

SUMMARY:
Maternal hypotension is a common problem during cesarian section under spinal anesthesia. The possible explanation for this is combined aortocaval compression by gravid uterus in parturient in addition to reduced systemic vascular resistance by spinal anesthesia. The investigators evaluated if the incidence of hypotension would be decreased by delayed supine positioning, by maintaining lateral position for 6 min after spinal injection, in patients undergoing elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* singleton parturients undergoing elective cesarean section
* gestational age over 37 weeks

Exclusion Criteria:

* pregnancy with hypotension
* expecting fetal depression

Ages: 28 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
hypotension | after intrathecal injection until delivery (for 20 minutes)
  hypotension incidence after intrathecal injection until baby delivery. Monitoring about for 20 minutes

SECONDARY OUTCOMES:
sensory block level | during cesarean section
  highest sensory block level after intrathecal injection